CLINICAL TRIAL: NCT02948764
Title: RESPONDER Trial - Diagnosis of Pathological Complete Response by Vacuum-assisted Biopsy After Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: Diagnosis of Pathological Complete Response by Vacuum-assisted Biopsy After Neoadjuvant Chemotherapy in Breast Cancer
Acronym: RESPONDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Jörg Heil, Prof. Dr. Joerg Heil, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2
Record Dates: First submitted 2016-10-16; First posted 2016-10-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; vacuum-assisted biopsy; pathological complete response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm study (Other): This project is designed as a one-armed diagnostic study. Every patient included in the study will undergo the same diagnostic test, the vacuum-assisted biopsy, after NACT and before surgery according to guidelines.
  Interventions: Device: Vacuum-Assisted Biopsy

INTERVENTIONS:
Device: Vacuum-Assisted Biopsy — The vacuum-assisted (7-10G), minimal invasive biopsy (VAB), either guided by ultrasound, or by mammography (stereotaxy) during the second trial visit (V2) will be performed once. In analogy to the German S3 guideline on primary breast cancer management we recommend to take at least 12 biopsies with 10G needles or less in case of larger needle sizes.
  Other Names: minimal invasive biopsy

SUMMARY:
The main purpose of the study is to evaluate the potential of a minimal invasive, vacuum-assisted biopsy (VAB) to reliably diagnose a pathological complete response (pCR) in the breast after neoadjuvant chemotherapy (NACT) in breast cancer patients.

The study is designed as a multicenter, confirmative, one-armed, intra-individually-controlled, open, diagnostic trial, in which we aim to confirm the applicability of preoperative VAB in patients after NACT. Furthermore, we aspire to quantify the rate of concordant pathological findings (pCR yes / no) in biopsy and surgical specimen.

DETAILED DESCRIPTION:
In clinical routine surgical treatment follows the pre-operative chemotherapy (NACT). However, recent studies have demonstrated that shrinking tumors need less surgical treatment indicating that patients with pCR could potentially be spared of surgery in the future. However, up to now, prediction of pCR after NACT is only moderately accurate. This prospective, monocenter diagnostic trial aims to explore if minimal invasive biopsies (MIB) might overcome this diagnostic challenge.

Ultrasound guided VAB will be performed on 600 breast cancer patients after NACT and directly prior to surgery.

There are only two trial visits that are specific to the trial. All other visits will be routine visits.

1. The first trial visit will take place in order to provide the patient with detailed information on the study, its' aims, the VAB procedure, and its risks. The patient will be asked to sign a form of informed consent.
2. At the second trial visit the performance of the VAB (=index test) will take place. This trial visit may vary by patient, tumor, and trial site characteristics and may either be:

   1. An ultrasound guided VAB or
   2. A stereotactically / mammographically guided VAB. All possible VAB procedures and settings (in outpatient clinic, or in operating room directly before the surgery) are equally accepted. We will allow every trial site to choose the adequate setting to the trial site´s and to their patients' needs.

A visit for a follow up will not be necessary in this setting. Possible complications of the VAB procedure may occur while the biopsy is taken.

The pathological results of the VAB specimen will be generally categorized as follows:

1. Residual tumor cells in VAB specimen (=non-pCR)
2. No residual tumor cells in the VAB specimen and VAB representative of former tumor region (="pCR in VAB")
3. No residual tumor cells in the VAB specimen but VAB unclear or not representative of former tumor region (=possible sampling error). These VABs are categorized as uninformative for the primary endpoint of the clinical trial.

The results will be compared to those of the pathological examination of surgical specimen.

ELIGIBILITY:
Inclusion Criteria

* Female patients with primary breast cancer after Neoadjuvant Chemotherapy (NACT) treatment which has been performed for at least 12 weeks and resulted in cPR or cCR (see below).
* >/=18 years
* any cT and cN stage, except cT4 stages
* any routine breast cancer surgical intervention planned according to guidelines (breast conservation or mastectomy)
* Residual intramammary target lesion or clip marker is visible in ultrasound and / or mammography
* Diagnosis of imaging complete or partial response according to RECIST 1.1 by at least mammography or ultrasound, according to local routine)
* Inclusion of only one breast per patient, in bilateral cancer one breast can be included
* In case of multicentric disease: confirmation of the same tumorbiological subtype defined by immunohistology in at least 2 lesions.
* Ability of subject to understand character and individual consequences of the clinical trial.
* Written informed consent (must be available before enrolment in the trial).

Exclusion Criteria

* Palliative or recurrent breast cancer
* in case of clip marker = target lesion: dislocation of marker (>5mm distance to the initial lesion border at the time of clip placement)
* contraindication for VAB or associated procedures (e.g. local anesthesia)
* Pregnancy and lactation
* held in an institution by legal or official order
* legally incapacitated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
false negative VAB results, reported as the false negative rate (= FNR) | after breast surgery, up to 6 weeks after VAB
  non-detected residual tumor by VAB (=index test) compared to breast surgery (=reference test): FNR = rate of patients with non-detected residual tumor by VAB compared to breast surgery Residual tumor is defined as a positive result; in surgical specimen as well as in VAB.

SECONDARY OUTCOMES:
negative predictive value (NPV) | after breast surgery, up to 6 weeks after VAB
  The negative predictive value (NPV) will be calculated as the quotient of the number of cases with pCR in VAB and in surgical specimen (= true negative result), divided by the total number of cases with pCR in VAB.
  Residual tumor is defined as a positive result; in surgical specimen as well as in VAB.
positive predictive value (PPV) | after breast surgery, up to 6 weeks after VAB
  The positive predictive value (PPV) will be calculated as the number of biopsies with detected residual tumor cells in VAB and surgery (= true positive results) divided by the number of all cases with residual tumor cells in the VAB.
  Residual tumor is defined as a positive result; in surgical specimen as well as in VAB.
false positive rate (FPR) | after breast surgery, up to 6 weeks after VAB
  FNR = rate of patients with falsely diagnosed residual tumor by VAB compared to breast surgery Residual tumor is defined as a positive result; in surgical specimen as well as in VAB.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Heil, Professor, Principal Investigator — University of Heidelberg University Breast Unit, Department of Gynecology
Locations (1):
- University Breast Unit, Department of Gynecology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Schaefgen B, Mati M, Sinn HP, Golatta M, Stieber A, Rauch G, Hennigs A, Richter H, Domschke C, Schuetz F, Sohn C, Schneeweiss A, Heil J. Can Routine Imaging After Neoadjuvant Chemotherapy in Breast Cancer Predict Pathologic Complete Response? Ann Surg Oncol. 2016 Mar;23(3):789-95. doi: 10.1245/s10434-015-4918-0. Epub 2015 Oct 14. PMID 26467456
- [Result] Heil J, Kummel S, Schaefgen B, Paepke S, Thomssen C, Rauch G, Ataseven B, Grosse R, Dreesmann V, Kuhn T, Loibl S, Blohmer JU, von Minckwitz G. Diagnosis of pathological complete response to neoadjuvant chemotherapy in breast cancer by minimal invasive biopsy techniques. Br J Cancer. 2015 Dec 1;113(11):1565-70. doi: 10.1038/bjc.2015.381. Epub 2015 Nov 10. PMID 26554654
- [Derived] Pfob A, Sidey-Gibbons C, Rauch G, Thomas B, Schaefgen B, Kuemmel S, Reimer T, Hahn M, Thill M, Blohmer JU, Hackmann J, Malter W, Bekes I, Friedrichs K, Wojcinski S, Joos S, Paepke S, Degenhardt T, Rom J, Rody A, van Mackelenbergh M, Banys-Paluchowski M, Grosse R, Reinisch M, Karsten M, Golatta M, Heil J. Intelligent Vacuum-Assisted Biopsy to Identify Breast Cancer Patients With Pathologic Complete Response (ypT0 and ypN0) After Neoadjuvant Systemic Treatment for Omission of Breast and Axillary Surgery. J Clin Oncol. 2022 Jun 10;40(17):1903-1915. doi: 10.1200/JCO.21.02439. Epub 2022 Feb 2. PMID 35108029
- [Derived] Pfob A, Sidey-Gibbons C, Lee HB, Tasoulis MK, Koelbel V, Golatta M, Rauch GM, Smith BD, Valero V, Han W, MacNeill F, Weber WP, Rauch G, Kuerer HM, Heil J. Identification of breast cancer patients with pathologic complete response in the breast after neoadjuvant systemic treatment by an intelligent vacuum-assisted biopsy. Eur J Cancer. 2021 Jan;143:134-146. doi: 10.1016/j.ejca.2020.11.006. Epub 2020 Dec 8. PMID 33307491
- [Derived] Heil J, Sinn P, Richter H, Pfob A, Schaefgen B, Hennigs A, Riedel F, Thomas B, Thill M, Hahn M, Blohmer JU, Kuemmel S, Karsten MM, Reinisch M, Hackmann J, Reimer T, Rauch G, Golatta M. RESPONDER - diagnosis of pathological complete response by vacuum-assisted biopsy after neoadjuvant chemotherapy in breast Cancer - a multicenter, confirmative, one-armed, intra-individually-controlled, open, diagnostic trial. BMC Cancer. 2018 Aug 25;18(1):851. doi: 10.1186/s12885-018-4760-4. PMID 30144818